CLINICAL TRIAL: NCT02544737
Title: A Phase II Study of Apatinib for Patients With Heavily Pretreated, Metastatic Esophageal Cancer.
Brief Title: Apatinib for Metastatic Esophageal Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Cancer Hospital (Other)
Responsible Party: Principal Investigator, Shixiu Wu, MD, Hangzhou Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH
Record Dates: First submitted 2015-09-06; First posted 2015-09-09 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Esophageal Cancer; Metastatic Esophageal Cancer; Apatinib
Keywords: Esophageal cancer; Metastatic esophageal cancer; Apatinib
MeSH Terms: conditions — Esophageal Neoplasms | interventions — apatinib

ARMS (1):
- Apatinib arm (Experimental): Patients with metastatic lesions of esophageal cancer after been treated with surgery or definitive chemoradiotherapy receiving Apatinib (850mg) daily over 4 weeks.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Patients with metastatic lesions of esophageal cancer after been treated with surgery or definitive chemoradiotherapy receiving Apatinib (850mg) daily over 4 weeks.

SUMMARY:
Patients with esophageal cancer that had metastatic lesions after been treated with surgery or definitive chemoradiotherapy are being asked to participate in this study.

Apatinib is a small-molecule vascular endothelial growth factors receptor (VEGFR) tyrosine kinase inhibitor, similar to vatalanib (PTK787), but with a binding affinity 10 times that of vatalanib or sorafenib.

The purpose of this study is to determine what effects apatinib has on metastatic esophageal cancer. These effects include whether apatinib could shrink the tumor or slow down its growth and what side effects apatinib will have on the tumor.

DETAILED DESCRIPTION:
The purpose of this study is to determine what effects apatinib has on metastatic esophageal cancer patients after been treated with surgery or definitive chemoradiotherapy. These effects include whether apatinib could shrink the tumor or slow down its growth and what side effects apatinib will have on the tumor.

Eligible are patients with metastatic esophageal cancer who have achieved stable disease or have disease progression after systemic therapy (surgery or definitive chemoradiotherapy) and have at least one separate measurable sites of metastatic lesions. Extent of metastatic disease is recorded either at CT or MRI scanning. Apatinib (850mg) is given daily during the therapy for 28 days. Tumor response is evaluated by assessing clinical and CT/MRI response in the metastatic sites. A Phase II clinical trial based on an optimum two-stage Phase II Simon design is used to conduct this pilot study. Ten patients will be treated in Stage one; if there are no tumor responses, the trial will be terminated. If there are one or more responses in Stage One, the trial will proceed to enroll an additional 19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed esophageal cancer which is persistent and metastatic or recurrent and metastatic;
2. Patients must have distinct measurable metastatic sites at least 1 cm of larger in their largest diameter;
3. Age ≥18 years;
4. Metastatic disease measurable on a CT/MRI scan. The primary tumor is not considered measurable disease. Metastatic lesions within a prior radiation field are acceptable as long as disease has progressed in the radiation field by RECIST criteria. The same imaging modality performed at baseline (CT or MRI) will be repeated at subsequent imaging.
5. ECOG performance status: 0-1;
6. Life expectancy ≥ 3 months.
7. Patients have adequate baseline organ and marrow function as defined by an absolute neutrophil count greater than 1500 cells per μL, platelet concentration of greater than 50 000 per μL, total bilirubin less than 1•5 times the upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase less than 2•5 times the ULN, and serum creatinine less than 1•5 times the ULN;
8. Signed consent forms voluntarily;

Exclusion Criteria:

1. Patients who have had prior allergic reaction to Apatinib;
2. Patients undergoing therapy with other investigational agents.
3. Women who are pregnant or breastfeeding;
4. Patients with known brain metastases can be included in this clinical trial but brain lesions are not eligible as target or non target lesion;
5. Anticipated patient survival under 3 months;
6. Active severe infection or known chronic infection with HIV, hepatitis B virus, or hepatitis C virus;
7. Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, myocardial infarction, stroke or congestive heart failure within the last 6 months;
8. The subject has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin;
9. Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities;
10. Patients with any other concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with response (CR, PR, SD and PD based on RECIST version 1.0) assessed at 5-6 weeks after the initiation of treatment. | week 5- week 6

SECONDARY OUTCOMES:
The number of participants with adverse events from the date of enrollment until 2 years from the opening of the study. | year 0- year 2
The proportion of patients alive (overall survival rate) from the date of enrollment until date of death from any cause, assessed up to 2 years from the opening of the study. | year 0- year 2

CONTACTS AND LOCATIONS:
Overall Officials: Shixiu Wu, MD, Study Chair — Hangzhou Cancer Hospital
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Golden EB, Chhabra A, Chachoua A, Adams S, Donach M, Fenton-Kerimian M, Friedman K, Ponzo F, Babb JS, Goldberg J, Demaria S, Formenti SC. Local radiotherapy and granulocyte-macrophage colony-stimulating factor to generate abscopal responses in patients with metastatic solid tumours: a proof-of-principle trial. Lancet Oncol. 2015 Jul;16(7):795-803. doi: 10.1016/S1470-2045(15)00054-6. Epub 2015 Jun 18. PMID 26095785
- [Background] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952